

# Device Protocol for CLY935-C019 / NCT04980456 Title: Clinical Assessment of Two Daily Wear Monthly Replacement Soft Silicone Hydrogel Contact Lenses

Protocol Number: CLY935-C019

Clinical Investigation

Type:

Postmarket Interventional / Confirmatory

Test Product: soft contact lenses (TOTAL30)

lehfilcon A

Sponsor Name and Alcon Research, LLC, and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Property of Alcon Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Alcon


Document ID: V-CLN-0010874

Status: Approved, Version: 1.0 Approved Date: 28 Jun 2021

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and
  agree to conduct the described trial in compliance with Good Clinical Practices;
  applicable international and national regulations, laws, guidelines, and standards; the
  conditions of approval imposed by the reviewing IRB or regulatory authority; and in
  accordance with the ethical medical research principles outlined in the Declaration
  of Helsinki.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as
  described in the protocol, current investigator's brochure, product information, or
  other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | | |
|---|---|---|---|---|
| | □ No | □Yes | | |
| | Have you | ever been | involved in a study or other resear | rch that was terminated? |
| | □ No | □Yes | | |
| | If yes, ple | ease explair | here: | |
| Pr | incipal inv | estigator: | | |
| | | | Signature | Date |
| | ame and pr<br>sition: | ofessional | | |
| Αc | ldress: | | | |
| Ph | one Numb | er: | | |
| | Off-hours Emergency<br>Phone Number: | | | |

# **Table of Contents**

| De | vice Proto | ocol for CLY935-C019 | 1 |
|---|---|---|---|
| Tal | ble of Cor | ntents | 3 |
| Lis | st of Table | S | 5 |
| Lis | st of Figur | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | ACRONYMS AND ABBREVIATIONS | 13 |
| 3 | PROTO | COL SUMMARY | 15 |
| 4 | PROTO | COL AMENDMENTS | 24 |
| 5 | INTROI | DUCTION | 24 |
| | 5.1 | Rationale and Background | 24 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | 25 |
| 6 | STUDY | OBJECTIVES | 26 |
| | 6.1 | Primary Objective(s) | 26 |
| | 6.2 | Secondary Objective(s) | 26 |
| | 6.4 | Safety Objective(s) | |
| 7 | INVEST | TIGATIONAL PLAN | 27 |
| | 7.1 | Study Design | 27 |
| | 7.2 | Rationale for Study Design | 28 |
| | | 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations | 20 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | |
| | 7.4 | Rationale for Choice of Comparator Product | |
| | 7.5 | Data Monitoring Committee | 29 |
| 8 | STUDY | POPULATION | 29 |
| | 8.1 | Inclusion Criteria | 30 |
| | 8.2 | Exclusion Criteria | 31 |
| | 8.3 | Rescreening of Subjects | 32 |
| 9 | TREATI | MENTS ADMINISTERED | 32 |

| | 9.1 | Investigational Product(s) | 32 |
|---|---|---|---|
| | 9.2 | Other Medical Device or Medication Specified for Use During the Study | y36 |
| | 9.3 | Treatment Assignment / Randomization | 37 |
| | 9.4 | Treatment masking | |
| | 9.5 | Accountability Procedures | 39 |
| | 9.6 | Changes to concomitant medications, treatments/ procedures | 40 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | 40 |
| | 10.1 | Informed Consent and Screening | 40 |
| | 10.2 | Description of Study Procedures and Assessments | |
| | | 10.2.1 Demographics | |
| | | 10.2.2 Medical History | |
| | | 10.2.3 Investigational Product compliance | 41 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 41 |
| | | 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment | 41 |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 42 |
| | | 10.2.7 Additional Study Assessments | |
| | 10.3 | Unscheduled Visits | 42 |
| | 10.4 | Discontinued Subjects | 42 |
| | | 10.4.1 Screen Failures | 42 |
| | | 10.4.2 Discontinuations | 43 |
| | | 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product | 43 |
| | 10.5 | Clinical Study Termination | 43 |
| | | 10.5.1 Follow-up of subjects after study participation has ended | 44 |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 44 |
| | 11.1 | General Information | 44 |
| | 11.2 | Monitoring for Adverse Events | 47 |
| | 11.3 | Procedures for Recording and Reporting | 47 |
| | 11.4 | Return product analysis, if applicable | 49 |
| | 11.5 | Unmasking of the Study Treatment | 49 |
| | 11.6 | Follow-Up of Subjects with Adverse Events | 50 |
| | 11.7 | Pregnancy in the Clinical Study | |
| 12 | | SIS PLAN | |
| | | Subject Evaluability | 51 |
| | 17.1 | DIDDING EVALUATION | ) I |

| 12.2 | Analysis Sets | 51 |
|-----------|----------------------------------------------------------|----|
| | 12.2.1 Safety Analysis Set | 51 |
| | 12.2.2 Full Analysis Set | 51 |
| 12.3 | Demographic and Baseline Characteristics | 51 |
| 12.4 | Effectiveness Analyses | 51 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 52 |
| | 12.4.1.1 Statistical Hypotheses | |
| | 12.4.1.2 Analysis Methods | 52 |
| 12.5 | Handling of Missing Data | 55 |
| 12.6 | Safety Analyses | 55 |
| 12.7 | Interim Analyses and Reporting | 56 |
| 12.8 | Sample Size Justification | |
| | ANDLING AND ADMINISTRATIVE REQUIREMENTS | |
| 13.1 | Subject Confidentiality | 58 |
| 13.2 | Completion of Source Documents and Case Report Forms | |
| 13.3 | Data Review and Clarifications | 59 |
| 13.4 | Sponsor and Monitoring Responsibilities | 59 |
| 13.5 | | |
| 13.6 | Quality Assurance and Quality Control | 60 |
| 14 ETHICS | | 60 |
| 15 REFERE | ENCES | 62 |
| 15.1 | Regulations and Standards | 62 |
| 16 APPENI | DIX A – Protocol Amendments | 62 |
| | T 2-4 - 6 T-11 | |
| Table 2 1 | List of Tables | 10 |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | 13 |
| Table 3–1 | Schedule of Study Procedures and Assessments | 21 |

| Document ID:<br>V-CLN-001087 | 4 | Status: Approved, Version: 1.0<br>Approved Date: 28 Jun 2021 | |
|---|---|---|---|
| Table 6–1 | Primary Objective(s) | | 26 |
| Table 6–3 | Safety Objective(s) | | 27 |
| Table 9–1 | Test Product | | 32 |
| Table 9–2 | Comparator Product | | 35 |
| | | List of Figures | |
| Figure 7-1 | Flowchart of Study Vis | sits | 28 |

Figure 11-1

Figure 11-2

# 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to as soft contact lenses or contact lenses |
|---|---|
| Name of Comparator<br>Product(s) | CooperVision® Biofinity® soft contact lenses (Biofinity) |
| Adverse Device Effect (ADE) | Adverse event related to the use of an investigational medical device (investigational product) or control product. Note: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation; any malfunction; and use error or intentional misuse of the investigational medical device (investigational product) or control product. |
| Adverse Event (AE) | Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (investigational product). Note: This definition includes events related to the investigational medical device, comparator, or the procedures involved. For users or other persons, this definition is restricted to events related to the use of investigational medical devices (investigational product) or control product. Requirements for reporting Adverse Events in the study can be found in Section 11. |
| Anticipated Serious Adverse Device Effect (ASADE) | An effect which by its nature, incidence, severity, or outcome has been identified in the risk assessment. |

| CILL II | |
|---|---|
| Clinical Investigation Plan | The document(s) stating the rationale, objectives, design, |
| (CIP) | and prespecified analysis, methodology, organization, |
| | monitoring, conduct, and record-keeping of the clinical |
| | investigation. |
| | Note: The protocol and other documents referenced in the |
| | protocol (for example, the Statistical Analysis Plan, the |
| | Manual of Procedures, the Deviations and Evaluability |
| | Plan, and the Protocol Monitoring Plan) comprise the CIP. |
| Clinical Investigation | The document describing the design, execution, statistical |
| Report (CIR) / Clinical | analysis, and results of a clinical investigation. The Clinical |
| Study Report | Investigation Report is synonymous with the Clinical Study |
| Study Report | Report. |
| | Report. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, |
| | quality, durability, reliability, usability, safety, or |
| | performance. |
| | Note: This definition includes malfunctions, use errors, and |
| | inadequacy in the information supplied by the manufacturer |
| | including labelling. |
| | Requirements for reporting Device Deficiencies in the study |
| | can be found in Section 11. |
| | Country of Total and Social Country of the Country |
| Enrolled Subject | Any subject who signs an informed consent form for |
| | participation in the study. |
| Point of Enrollment | The time at which, following recruitment and before any |
| | clinical investigation-related procedures are undertaken, a |
| | subject signs and dates the informed consent form. |
| Interventional Clinical Trial | A pre- or postmarket clinical investigation where the |
| interventional Chinear IIIai | assignment of a subject to a particular medical device is |
| | decided in advance by a clinical investigation plan, or |
| | diagnostic or monitoring procedures requested in the CIP are |
| | in addition to those available as normal clinical practice and |
| | burden the subject. |

| Investigational Product | A preventative (vaccine), a therapeutic (drug or biologic), device, diagnostic, or palliative used as a test or comparator product in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized form. |
|---|---|
| Malfunction | Failure of an investigational medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or clinical investigation plan (CIP), or investigator's brochure (IB). |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |
| Product Complaint | Any oral, electronic, or written communication that alleges deficiencies related to the identity (labeling), quality, durability, reliability, safety, effectiveness, or performance of a marketed product, including failure of the product, labeling, or packaging to meet specifications, whether or not the product is related to or caused the alleged deficiency. A complaint may allege that an adverse event or medical device malfunction has occurred. |
| Randomized Subject | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device<br>Effect (SADE) | Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event. |

# Serious Adverse Event (SAE)

Adverse event that led to any of the following:

- Death.
- A serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - a) a life-threatening illness or injury

    Note: Life-threatening means that the individual was
    at immediate risk of death from the event as it
    occurred, i.e., it does not include an event which
    hypothetically might have caused death had it
    occurred in a more severe form.
  - any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases.
  - c) inpatient hospitalization or prolonged hospitalization.

Note: Planned hospitalization for a preexisting condition, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an outpatient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

- d) a medical or surgical intervention to prevent a) or b).
- e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.

| | Fetal distress, fetal death, congenital abnormality or birth defect including physical or mental impairment. Note: Planned hospitalization for a preexisting condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event. |
|---|---|
| | Refer to Section 11 for additional SAEs. |
| Serious Health Threat | Signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users, or other persons, and that requires prompt remedial action for other subjects, users, or other persons. |
| | Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
| Significant Nonserious | A symptomatic, device-related, non-sight-threatening |
| Adverse Event | adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. |
| | Refer to Section 11 for additional Significant Nonserious AEs. |
| Study Start | The start of the study is considered to coincide with the enrollment of the first patient. |
| Study Completion | The completion of the study is considered to coincide with<br>the study-level last subject last visit or the decision to<br>terminate the trial, whichever is later. |
| Unanticipated Serious<br>Adverse Device Effect<br>(USADE) | Serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the risk assessment. |

| Use Error | User action or lack of user action while using the medical |
|---|---|
| | device that leads to a different result than that intended by |
| | the manufacturer or expected by the user. |
| | Note: |
| | a) Use error includes the inability of the user to complete a task. |
| | b) Use errors can result from a mismatch between the characteristics of the user, user interface, task, or use environment. |
| | c) Users might be aware or unaware that a use error has occurred. |
| | d) An unexpected physiological response of the patient |
| | is not by itself considered a use error. |
| | e) A malfunction of a medical device that causes an |
| | unexpected result is not considered a use error." |

### 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2-1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| ASADE | Anticipated serious adverse device effect |
| BCVA | Best corrected visual acuity |
| Biofinity | CooperVision Biofinity soft contact lenses (Biofinity) |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CIP | Clinical investigation plan |
| CIR | Clinical investigation report |
| CLEAR CARE | CLEAR CARE® Cleaning & Disinfecting Solution |
| COL | Clinical Operations Lead |
| CRF | Case report form |
| CSM | Clinical Site Manager |
| D | Diopter(s) |
| DEP | Deviations and evaluability plan |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EN | European Standard |
| FAS | Full analysis set |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LacriPure | Menicon LacriPure, Rinsing & Insertion Saline, Preservative free |
| | saline |
| LogMAR | Logarithm of the minimum angle of resolution |
| MOP | Manual of procedures |
| N | Number of subjects |
| NI | Noninferiority |
| OD | Right eye |
| OS | Left eye |

| Abbreviation | Definition |
|--------------|---------------------------------------------|
| PHXB6 | PHXB6 core material |
| PP | Per protocol |
| R&D | Research & Development |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SD | Standard deviation |
| Seq | Sequence |
| SLE | Slit lamp examination |
| SOP | Standard operating procedure |
| US | United States |
| USADE | Unanticipated serious adverse device effect |
| USV | Unscheduled visit |
| VA | Visual acuity |

# 3 PROTOCOL SUMMARY

| Investigational | Device |
|---|---|
| product type | |
| Study type | Interventional |
| Investigational | Test Product: |
| products | Comparator Product: CooperVision Biofinity soft contact lenses (Biofinity) |
| Purpose and | To compare the clinical performance of contact lenses |
| Scientific Rationale | with Biofinity contact lenses over 30 days of daily wear |
| for the Study | |
| Objective(s) | The <b>primary objective</b> of this study is to demonstrate |
| | noninferiority (NI) in visual acuity at distance when wearing |
| | contact lenses compared to Biofinity contact lenses. |
| Endpoint(s) | Primary effectiveness |
| | Distance VA (logMAR) with study lenses at Day 30 |





| Sites and Locations | Planned number of subjects enrolled/consented: ~260 Planned number of completed subjects: 232 Planned number of clinical sites: 12-16 Planned locations (initial list of locations, which may change during start up or conduct according to study needs): US |
|---|---|
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Current wearers of any commercial spherical weekly/monthly soft contact lenses with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.</li> <li>Manifest cylinder ≤ 0.75 D in each eye.</li> <li>Best corrected distance visual acuity better than or equal to 20/25 Snellen in each eye (as determined by manifest refraction at screening).</li> </ul> |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | <ul> <li>Monovision or multifocal lens wearers.</li> <li>Habitual Biofinity contact lens wearers (in the past 3 months).</li> <li>Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.</li> </ul> |





Table 3-1 Schedule of Study Procedures and Assessments

| | | Lens 1<br>(Period 1) | | Lens 2<br>(Period 2) | | | |
|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | Prescreening | Visit 1 Screen/ Baseline/ Dispense Lens 1 [Day 1] | Visit 2 Follow-up Lens 1 [Day 30 ± 2 days] | Visit 3 Dispense Lens 2 [Day 1] | Visit 4 Follow-up Lens 2 / Exit [Day 30 ± 2 days] | Early<br>Exit | usv |
| Informed Consent | | X | | | | | |
| Demographics | | X | | | | | |
| Medical History <sup>¥</sup> | | X | X | X | X | X | X |
| Concomitant Medications* | | X | X | X | X | X | X |
| Pregnancy | | X | X | X | X | X | X |
| Inclusion/ Exclusion | | X | | | | | |
| Habitual (lens brand, lens power*, lens care) | | X | | | | | |
| VA w/ habitual correction* (OD, OS, Snellen distance) | | X | | | X | X | (X) |
| Manifest Refraction and BCVA with manifest refraction* (OD, OS, Snellen distance) | | X | (X) | (X) | (X) | (X) | (X) |
| Biomicroscopy | | X | X | X | X | X | (X) |
| Randomization and record lens power* | | X | | | | | |
| Dispense study lenses | | X | | X | | | (X) |
| VA w/ study lenses (OD, OS, logMAR distance) | | X | X | X | X | X | (X) |


| | pn | Lens<br>(Perio | | | ens 2<br>riod 2) | | |
|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | Prescreening | Visit 1 Screen/ Baseline/ Dispense Lens 1 [Day 1] | Visit 2 Follow-up Lens 1 [Day 30 ± 2 days] | Visit 3<br>Dispense<br>Lens 2<br>[Day 1] | Visit 4 Follow-up Lens 2 / Exit [Day 30 ± 2 days] | Early<br>Exit | USV |
| Collect worn lenses* <sup>β</sup> | | | X | | X | X | (X) |
| AEs§ | | X | X | X | X | X | X |
| Device deficiencies | | X | X | X | X | X | X |
| Exit Form | | | | | X | X | |

USV = Unscheduled visit; EOD = End of Day

\* Source only

#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 5 INTRODUCTION

#### 5.1 Rationale and Background

Daily wear contact lenses are worn during waking hours, often for a full day and then removed for cleaning and disinfection prior to reinsertion the following day. Frequent replacement daily wear contact lenses are replaced according to the product package insert provided by the contact lens manufacturer.

New silicone hydrogel materials continue to be developed, possessing unique material properties and superior oxygen transmissibility over contact lenses made with conventional hydrogel materials. A new lens, known as the contact lens, has been developed in an effort to maintain sustained performance by providing an inherently wettable core material with a water gradient surface. The new silicone hydrogel lens has been designed to provide favorable performance for daily wear with 1-month replacement.

In this clinical study, the clinical performance of the investigational contact lens will be assessed and the contact lens will be compared to the commercially available Biofinity contact lens in a crossover design, both to be worn in a daily wear modality for approximately 1 month.

# 5.2 Purpose of the Study

| The purpose of this study is to assess the clinical performance of the investigational |
|---|
| contact lens over 30 days of daily wear compared to Biofinity. The primary endpoint was |
| selected to address the primary objective of the study. |
| The design of this |

study is justified based upon preclinical and clinical testing, as described within the Investigator's Brochure. Biofinity contact lenses were chosen as the comparator product because these lenses have the same wear modality and replacement schedule.

At the end of the study, a clinical study report will be prepared in accordance with applicable regulatory requirements and standards.



#### 5.3 Risks and Benefits

The clinical investigation process risks are managed through appropriate training and monitoring according to the protocol-specific monitoring plan. Investigational device risks, including risks associated with use of device and methods and procedures for application of device, are defined in the investigator's brochure and/or product labeling and are managed through review of safety assessments outlined in this protocol.

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of contact lenses are features consistent with successful contact lens wear. Based upon nonclinical testing and documented rationale for applicability of test results, contact lenses are assessed to be nontoxic and biocompatible for on-eye use.

In the US, Biofinity contact lenses have approved indications for use for both daily wear and extended wear for up to 6 continuous nights. Further details on any known potential risks and benefits can be found in the product package insert.

There may also be unknown risks to use of contact lenses. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight and monitoring.

Refer to the IB for additional information.

### 6 STUDY OBJECTIVES

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Demonstrate noninferiority in VA at | Distance VA (OD, OS; logMAR) at Day 30 |
| distance when wearing contact | |
| lenses compared to Biofinity contact lenses. | |

# 6.2 Secondary Objective(s)

Not Applicable





# 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the study products | <ul><li>Adverse events</li><li>Biomicroscopy findings</li></ul> |
| | Device deficiencies |

# 7 INVESTIGATIONAL PLAN

#### 7.1 Study Design

| 7.1 Study Design |
|---|
| This is a prospective, interventional, randomized, double-masked, bilateral crossover study evaluating visual acuity of the investigational contact lens. Habitual spherical |
| weekly/monthly soft contact lens wearers |
| will be randomized in 1 of the 2 crossover sequences. |
| Subjects and investigators will be masked. An unmasked study staff member will prepare the contact lenses for dispensing. |
| Subjects will be expected to attend 4 office visits. All study contact lenses will be prescribed according to subject's prescription. CLEAR CARE contact lens solution will be used for daily contact lens cleaning and disinfection. |
| Subjects will be expected to wear the study contact lenses every day for at least 10 hours per day over a 30 day period per study lens. |

The total expected duration of a subject's participation is approximately 65 days,

The study is expected to be completed in approximately 3 months.

Figure 7-1 Flowchart of Study Visits



# 7.2 Rationale for Study Design

This study design is justified based upon an evaluation of the results of relevant preclinical and clinical testing, as described within the IB.

The crossover design will ensure that the same subject is exposed to both the test and comparator lens materials;

The study will include only those subjects who are current wearers of spherical weekly/monthly soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day. This will avoid confounding safety responses in nonadapted subjects. Furthermore, the subjects will not be permitted to use lubrication/rewetting drops during lens wear as this may confound the primary effectiveness endpoint. However, habitual lubrication/rewetting drops usage is allowed prior to lens insertion and after lens removal. No lubrication/rewetting drop use allowed during clinic visits.

The study will exclude any habitual Biofinity contact lens wearers in the past 3 months prior to consent in order to reduce potential bias of wearers to their habitual contact lenses. The study will also exclude subjects who are monovision or multifocal contact lens wearers.

# 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations

An interim analysis will not be performed.

#### 7.3 Rationale for Duration of Treatment/Follow-Up

Subjects will wear each study product bilaterally for approximately 30 days, which represents the planned replacement period for both products. The lenses will be provided by a qualified unmasked study staff member in such a manner that the subject and the investigator remain masked to the lens type.

#### 7.4 Rationale for Choice of Comparator Product

Biofinity contact lenses were chosen as the comparator product because these lenses have the same wear modality and replacement schedule.

## 7.5 Data Monitoring Committee

Not applicable.

#### 8 STUDY POPULATION

The study population consists of male and female subjects aged 18 years or older who are current wearers of spherical weekly/monthly soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.

This study aims to enroll (consent) approximately 260 subjects in 12-16 US sites, with a target of 245 randomized, with 14 (intended minimum) to 25 (intended maximum) subjects per site. Additional subjects may be enrolled at specific sites with prior sponsor approval. Site-specific targets may vary based upon individual site capabilities. Estimated time needed to recruit subjects for the study is approximately 6 weeks;

however, unanticipated circumstances may shorten or lengthen this time and would not require amendment of this protocol.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- Subjects must be able to understand and sign an IRB/IEC approved Informed Consent form.
- 2. Subjects must be  $\geq$  18 years of age.
- 3. Willing and able to attend all scheduled study visits as required per protocol.
- 4. Current wearers of a commercial spherical weekly/monthly soft contact lenses with at least 3 months wearing experience prior to enrollment, with a minimum wearing time of 5 days per week and 10 hours per day.
- 5. Manifest cylinder  $\leq 0.75$  D in each eye.
- 6. Able to wear contact lenses within a range of sphere power from -1.00 to -6.00 D (0.25 D steps) and subject willing and able to wear the study lenses every day for at least 10 hours per day for the full duration of the study
  9. Subjects must be willing to stop wearing their habitual contact lenses for the duration of study participation.

#### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

- 1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.



4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study.



- 10. Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear, during the study.



14. Habitual comfilcon A (e.g., Biofinity, Biofinity Energys) contact lens wearers (in the past 3 months, prior to screening).

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be documented on the applicable eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis. Moreover, subjects who become pregnant during the study will not be discontinued; however, data will be excluded from the effectiveness analyses because pregnancy can alter refraction and visual acuity results.

### 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

#### 9.1 Investigational Product(s)

Test Product(s):

Comparator Product(s) (If CooperVision Biofinity soft contact lenses (Biofinity) applicable):

Table 9–1 Test Product

| Test Product | The lehfilcon A lenses received FDA 510(k) clearance on April 12, 2021 |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway |

| | Fort Worth, Texas 76134-2099 |
|---|---|
| | USA |
| Indication for use | The intended use of this product is for vision correction. |
| and intended | |
| purpose in the | |
| current study | |
| Product description | Material: lehfilcon A, |
| and parameters | • Water content: $55\% \pm 2\%$ |
| available for this | • Power range: -1.00 to -6.00 D (0.25 D steps) |
| study | Base curve (mm): 8.4 |
| | • Diameter (mm): 14.2 |
| Usage | Wear: |
| | o Daily Wear |
| | o Bilateral |
| | <ul> <li>Crossover according to randomization</li> </ul> |
| | Replacement period: Replacement lenses will not be provided to |
| | the subject. In the event a lens needs to be replaced, the subject |
| | must return to the site for a replacement lens. |
| | · |
| | Exposure: At least 10 hours per day, every day, over a 30-day |
| | period. |
| | Lens Care: Cleaned and disinfected with CLEAR CARE |
| | LacriPure or equivalent will be permitted for rinsing the lenses |
| | after removal or prior to insertion (as needed) |
| | Lubrication/rewetting drops will not be permitted during lens |
| | wear. However, habitual lubrication/rewetting drops usage is |
| | allowed prior to lens insertion and after lens removal. No |
| | lubrication/rewetting drop use allowed during clinic visits. |
| | Instructions for use will be provided in a separate document |

| Number/Amount of | Subjects will insert study lenses at Visit 1 and Visit 3 at the site. No |
|---|---|
| product to be | spare lenses will be provided to the subject. |
| provided to the | |
| subject | |
| Packaging | Blister foil pack |
| description | |
| Labeling description | Lens Foil label includes: |
| | - identifier |
| | - base curve |
| | - diameter |
| | - manufacturing protocol number |
| | - packing solution |
| | - power |
| | - lot number |
| | - expiration date |
| | - content statement |
| | <ul> <li>investigational device statement</li> </ul> |
| | - sponsor information |
| | - country of origin |
| | Provided in cartons of approximately 25 lenses per power, |
| | identified with the following: |
| | - a color coded label stating the protocol number |
| | - material identifier |
| | - power |
| | - an investigational device statement |
| m · | - handling unit |
| Training and/or | No additional training or experience is required to administer the |
| experience | test product. |
| requirements for | |
| device | |
| Storage conditions | Lens to be stored at room temperature. |
| Additional | An unmasked staff member will remove the contact lens from the |
| information | blister foil to preserve masking. |

| Supply | Alcon will provide an inventory of study lenses in each power. This |
|---|---|
| | inventory will be used for both fitting and subject lenses. Resupply |
| | of investigational product will be available upon request. |
| | CLEAR CARE contact lens solution, a contact lens case, and |
| | LacriPure (or equivalent) will be provided to the subject. |

Table 9–2 Comparator Product

| Comparator | Biofinity |
|---|---|
| Product(s) | (Not Biofinity Energys) |
| Manufacturer | CooperVision |
| Indication for Use | The intended use of this product is for vision correction. |
| Product description | Material: comfilcon A |
| and parameters | Water content: 48% |
| available for this | • Power range: -1.00 to -6.00 D (0.25 D steps) |
| study | Base curve (mm): 8.6 |
| | • Diameter (mm): 14.0 |
| Formulation | Silicone Hydrogel. For additional details, please refer to the |
| | Biofinity package insert. |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> <li>Crossover according to randomization</li> </ul> </li> </ul> |
| | Replacement period: Replacement lenses will not be provided to the subject. In the event a lens needs to be replaced, the subject must return to the site for a replacement lens. |
| | Exposure: At least 10 hours per day, every day, over a 30-day period. |
| | Lens Care: Cleaned and disinfected with CLEAR CARE |
| | LacriPure or equivalent will be permitted for rinsing the lenses after removal or prior to insertion (as needed) |

| Number/Amount of Product to be | <ul> <li>Lubrication/rewetting drops will not be permitted during lens wear. However, habitual lubrication/rewetting drops usage is allowed prior to lens insertion and after lens removal. No lubrication/rewetting drop use allowed during clinic visits.</li> <li>Instructions for use will be provided in a separate document</li> <li>Subjects will insert study lenses at Visit 1 and Visit 3 at the site. No spare lenses will be provided to the subject.</li> </ul> |
|---|---|
| Provided to the | |
| subject | |
| Packaging | Blister foil pack in commercial packaging. |
| description | |
| description | |
| Labeling description | Commercial labeling |
| Training and/or | No additional training or experience is required to administer the |
| experience | test product. |
| requirements for | |
| device | |
| Storage conditions | Lens to be stored at room temperature. |
| Additional | An unmasked staff member will remove the contact lens from the |
| information | blister foil to preserve masking. |
| Supply | Each site will procure their own comparator lenses. |
| | CLEAR CARE contact lens solution, a contact lens case, and LacriPure (or equivalent) will be provided to the subject. |

More information on the test product can be found in the investigator's brochure; information on the comparator product can be found in the Biofinity Package Insert.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

During the clinical study, the following contact lens solution is required in conjunction both study lenses:
- CLEAR CARE Cleaning & Disinfecting Solution
- LacriPure or equivalent will be permitted for rinsing the lenses after removal or prior to insertion (as needed)

Lubrication/rewetting drops will not be permitted during lens wear. However, habitual lubrication/rewetting drops usage is allowed prior to lens insertion and after lens removal. No lubrication/rewetting drop use allowed during clinic visits.

No other medical devices or medications are required to be used in conjunction with the treatments during the clinical study.

# 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 ratio to receive treatment in crossover sequence of Test product then Comparator product or Comparator product then Test product, respectively.

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment arms to randomization numbers in the specified ratio. Subjects will be assigned treatment according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/randomization integration to one of the treatment arms. The investigator's delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but will not be communicated to the site user. The EDC/randomization integration system will inform the site user of the treatment sequence (lens sequence) assignment to be dispensed to the subject.

# 9.4 Treatment masking





This level of masking will be maintained throughout the conduct of the study. Unmasking

This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

In the event of a medical emergency where the knowledge of subject treatment is required, an individual investigator will have the ability to unmask the treatment assignment for a specific subject after contacting an appropriate study sponsor representative if time allows.

## 9.5 Accountability Procedures

Upon receipt of the IPs, the investigator or delegate must conduct an inventory. During the study, the masked investigator must designate unmasked study staff to provide the IPs to the subjects in accordance with their randomization assignment. Throughout the study, the investigator or delegate must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the investigator must be accounted for by study sponsor personnel, and in no case be used in an unauthorized situation.

The investigator should make every effort to collect unused lenses, foils, and supplies from subjects.

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed

 Any study lenses associated with a device deficiency or with any product-related adverse event (i.e., ADE or SADE) are returned to the study sponsor for investigation, unless otherwise directed by the sponsor. Refer to Section 11 of this protocol for additional information on the reporting of device deficiencies and AEs and the return of study products associated with these events.

The investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

#### 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions).

The investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

#### 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

The investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

Prescreening for eligibility of potential subjects must be done the using the IRB-approved telephone prescreening script

#### 10.2 Description of Study Procedures and Assessments

Study-specific procedures and assessments described here may include standard of care; other standard of care procedures performed in the clinical management of the subject are not excluded.

Detailed descriptions of assessments and procedures are provided in the MOP. All study procedures and assessments are to be performed according to the table of procedures (Table 3-1). The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

#### 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

#### **10.2.2 Medical History**

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

Medical History and Concomitant Medications will be collected in the eCRF as outlined in the MOP.

# 10.2.3 Investigational Product compliance

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

# 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported since the previous visit, including those associated with changes in concomitant medication dosing. See Section 11 for further details regarding AE collection and reporting.

# 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber and lens must be performed in both eyes before instillation of any diagnostic eye drops.

#### 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any Device Deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11. Device deficiencies on comparator lenses should be reported per the manufacturer's guidelines.

### 10.2.7 Additional Study Assessments

Additional effectiveness assessments will be conducted throughout the course of the study. Refer to the MOP and Table 3-1 for details on each of these assessments.

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visit and the visit is conducted by study personnel, this visit must be documented as an Unscheduled Visit. If the subject seeks medical attention outside the clinic (for example, at an Emergency Room) or at the clinic but is seen by nonstudy personnel, the investigator is to capture adverse event-related information on the Adverse Event form upon becoming aware.

During all unscheduled visits, the investigator must conduct the following procedures:

- Collect Adverse Event information
- Collect device deficiency information
- Record changes in medical condition or concomitant medication

The investigator may perform additional procedures for proper diagnosis and treatment of the subject according to Table 3-1. The investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, as possible.

## 10.4 Discontinued Subjects

#### 10.4.1 Screen Failures

Subjects who were excluded from the study after signing the informed consent and prior to randomization to product/dispense of study product.

The investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing informed consent.

Subject numbers of discontinued subjects must not be re-used (i.e., subject replacement is not allowed).

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments, if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3-1.

## 10.5 Clinical Study Termination

The study sponsor reserves the right to suspend or close the investigational site or suspend or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the study sponsor:

• The study sponsor must:

- Immediately notify the investigator(s) and subsequently provide instructions for study termination.
- Inform the investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for poststudy treatment options as needed.

The investigator may terminate the site's participation in the study for reasonable cause.

Breaking of the masked treatment codes will be done after locking the database.

### 10.5.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All Adverse Events



Figure 11-2 Categorization of All Serious Adverse Events



#### Serious Adverse Events

In addition to reporting all AEs (serious and nonserious) meeting the definitions, the investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - Infiltrates > 2 mm diameter
  - Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon
- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting ≥ 50% of corneal surface area

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color)
- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack

- Packaging deficit (e.g., mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination
- Lack of performance

## 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

In addition, changes in any *protocol-specific parameters and/or questionnaires* evaluated during the study are to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in a *protocol-specific parameter or questionnaire response* that is clinically relevant, in the opinion of the investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

#### 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent Any preexisting medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the investigator must document all device deficiencies reported or observed with test and comparator products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

 All SAEs must be reported immediately (within 24 hours) of the investigator's or site's awareness.

- ADEs that do not meet seriousness criteria and device deficiencies must be reported within 10 calendar days of the investigator's or site's awareness.
- A printed copy of the completed Serious Adverse Event and Adverse Device Effect and/or Device Deficiency eCRF must be included with product returns
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
  Certificate of Death, etc., if applicable, in narrative section of the Adverse Device
  Effect (for related AEs) and Serious Adverse Event eCRF.

Note: Should the EDC system become nonoperational, the site must complete the appropriate paper Serious Adverse Event and Adverse Device Effect and/or Device Deficiency Form. The completed form is emailed to the study sponsor at msus.safety@Alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Any AEs and device deficiencies for nonstudy marketed devices/products (i.e. CLEAR CARE Cleaning & Disinfecting Solution, LacriPure (or equivalent)) will be considered and processed as spontaneous (following the postmarket vigilance procedures) and should be communicated to the device's/product's manufacturer as per local requirements.

Study sponsor representatives may be contacted for any protocol related question and their contact information is provided in the Manual of Procedures that accompanies this protocol.

Further, depending upon the nature of the AE or device deficiency being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

Intensity (Severity)


Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by study sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (i.e., there are other more likely causes for the AE).

The study sponsor will assess the AEs and may upgrade the investigator's assessment of seriousness and/or causality. The study sponsor will notify the investigator of any AEs that is upgraded from nonserious to serious or from unrelated to related.

# 11.4 Return product analysis, if applicable

Study sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

Alcon study products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint # which will be provided by study sponsor after the case is entered in the study sponsor's Global Product Complaint Management System (GPCMS).

# 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study (see Section 9.4). If the treatment code needs to be broken in the interest of

subject safety, the investigator is encouraged to contact an appropriate study sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (i.e., medical emergency), the code may be broken prior to contact with the study sponsor. The study sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the study sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

#### 11.6 Follow-Up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The investigator should provide the study sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of discontinuation, any additional information received at follow-up should be documented in the eCRFs up to study completion (i.e., database lock). Any additional data received up to 3 months after subject completed the study should be documented and available upon the study sponsor's request.

All complaints received after this time period will be considered and processed as spontaneous (following the postmarket vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements. The investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

# 11.7 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the appropriate eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case—by-case basis.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or

confidence limits where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

# 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens sequence) assignment and locking the database, based upon the deviations and evaluability plan (DEP).

#### 12.2 Analysis Sets

## 12.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

## 12.2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study.

# 12.3 Demographic and Baseline Characteristics

Demographic information will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, race, and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

# 12.4 Effectiveness Analyses

This study defines 1 primary, endpoint

The primary effectiveness endpoint of distance VA will be tested at one-sided  $\alpha$ =0.05 for noninferiority

## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate noninferiority in VA at distance when wearing contact lenses compared to Biofinity contact lenses. The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.

## 12.4.1.1 Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

 $H_0: \mu_{(T)} - \mu_{(C)} \ge 0.05$  $H_a$ :  $\mu_{(T)} - \mu_{(C)} < 0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for and Biofinity, respectively, on the logMAR scale.

# 12.4.1.2 Analysis Methods

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, visit, lens by visit interaction, period, and sequence. Withinsubject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference minus Biofinity) and the corresponding one-sided 95% upper confidence limit will be computed. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.







# 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary

# 12.6 Safety Analyses

The safety endpoints are:

- AEs
- · Biomicroscopy findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (frequencies and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation, significant nonserious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure) to any subsequent visit within the same period will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits within the same period for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure to study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be conducted for the safety analyses.

# 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.



Document ID: Status: Approved, Version: 1.0 V-CLN-0010874 Approved Date: 28 Jun 2021

## 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

## 13.1 Subject Confidentiality

The investigator must ensure that the subject's identity is kept confidential throughout the course of the study. In particular, the investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. The study sponsor may collect a copy of the enrollment log without any directly identifying subject information.

The study sponsor may share patient-level data collected in this trial with qualified researchers to help facilitate product development or enhancements in research that is not directly related to the study objectives. The Informed Consent explains this to the study subject.

#### 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study

Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The principal investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

#### 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will select principal investigators that are qualified by education, training, and experience to assume responsibility for the proper conduct of this clinical trial.

The study sponsor is financially funding this clinical trial and will compensate the investigator and/or the Institution(s) at which the study is conducted in accordance with a signed clinical trial agreement.

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate study sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written

and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

A coordinating investigator may be identified by the study sponsor to review and endorse the final study report. In cases where a coordinating investigator is engaged, the study sponsor will select the coordinating investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

#### 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the study sponsor. If the investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the study sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

## 13.6 Quality Assurance and Quality Control

The study sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the study sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the study sponsor with the investigator/institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

Investigations are conducted in compliance with Good Clinical Practices; international and national regulations, laws and guidelines; the conditions of approval imposed by reviewing IRBs/IECs or regulatory authorities; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.

 The SOPs of the study sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations shall apply.

 Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements.

The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The investigator must provide documentation of the IRB/IEC approval to the study sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the IB, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. At the end of the study, the investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject. The obtaining of consent shall be documented before any procedure specific to the clinical investigation is applied to the subject.

The investigator must have a defined process for obtaining the required consent. Specifically, the investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the investigator, and if required by local regulation, other qualified personnel. The investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate

individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and sponsor-designated personnel. The investigator must keep the original, signed copy of the consent (file in subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The study sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov if required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome if required by current regulations and, if applicable, in other public databases as required by local country regulations.

#### 15 REFERENCES

## 15.1 Regulations and Standards

The following references may be applicable in whole or in part for this clinical trial.

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- EN ISO 14155:2020 Clinical investigation of medical devices for human subjects -Good Clinical Practice
- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights, if applicable

#### 16 APPENDIX A – Protocol Amendments

There are no amendments. This is the first version of the protocol.

